CLINICAL TRIAL: NCT04733456
Title: Evaluation of Brain Activity and Oxygenation Using Near-infrared Spectroscopy (NIRS) in Inflammatory Bowel Disease (IBD) Patients
Brief Title: Brain Activity and Oxygenation Inflammatory Bowel Disease (IBD) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB20-1873
Record Dates: First submitted 2020-11-23; First posted 2021-02-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-11

CONDITIONS: IBD; Maladaptive Behavior Associated With Physical Illness
MeSH Terms: interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, stool and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD Patients (UC and CD): Participants will complete a Mayo Clinic Score (UC) or HBI score (CD), short IBDQ73, *EQ5D-5L, *GAD-774, *PHQ-975, *PROMIS (Gastrointestinal Belly Pain), Multidimensional Assessment of Interoceptive Awareness (MAIA)77, *Pain Catastrophizing Scale, Pittsburg Sleep Quality Index (PSQI) and Fatigue Severity Scale (FSS) at baseline and 16 weeks after the start of anti-TNF therapy (*questionnaires available through the CIHR IMAGINE grant).
  Stool will be collected at baseline and after 16 weeks for assessment of the known biomarker fecal calprotectin, in addition to fecal bacterial and fungal microbiome (through the International Microbiome Center [IMC], U of C). Blood will be drawn and urine collected at baseline and after 16 weeks for inflammatory markers and metabolomic [IMC] analysis
  Interventions: Behavioral: Quality of life questionnaires; Device: NIRS; Other: Stool Collection; Other: Blood and urine collection

INTERVENTIONS:
Behavioral: Quality of life questionnaires — Mayo Clinic Score (UC) or HBI score (CD), short IBDQ73, *EQ5D-5L, *GAD-774, *PHQ-975, *PROMIS (Gastrointestinal Belly Pain), Multidimensional Assessment of Interoceptive Awareness (MAIA)77, *Pain Catastrophizing Scale, Pittsburg Sleep Quality Index (PSQI) and Fatigue Severity Scale (FSS) at baseline and 16 weeks after the start of anti-TNF therapy
Device: NIRS — A TechEn NIRSOptix continuous-wave fNIRS system will be used to record changes in cerebral oxygenation, at a sampling rate of 25 Hz
Other: Stool Collection — For assessment of the known biomarker fecal calprotectin, in addition to fecal bacterial and fungal microbiome
Other: Blood and urine collection — for inflammatory markers and metabolomic [IMC] analysis

SUMMARY:
Symptoms such as fatigue, sleep disturbances, anxiety and depression are common in patients with IBD, but the cause is unknown. Understanding how these behaviors occur in IBD and their role in symptoms may help improve management of IBD. How IBD leads to changes in brain function remains unclear. Inflammation and dysfunction of blood flow may occur in patients with IBD, which may be linked to these symptoms. Patients with IBD also have an alteration or imbalance of gut bacteria which may play a role in the development of the disease, but the exact mechanism remains poorly understood;as a result, there are limited therapeutic options available clinically to address this issue. An approved therapy, anti-TNF α, may be useful in improving brain and gut activity as well as quality of life. The purpose of this research study is to better understand brain and gut activity in the context of IBD to possibly improve treatments for the disease. In patients taking anti-TNFα therapy as prescribed clinically as standard of care, the investigators will measure brain activity using NIRS; gut microbiome using stool analysis and quality of life using various questionnaires.

DETAILED DESCRIPTION:
Hypothesis Conditions with acute systemic inflammation will correlate with changes in gut microbiome signatures, reduced cerebral oxygen saturation (StO2) and altered patterns of microvascular cerebral blood perfusion (as determined by near-infrared spectroscopy NIRS).

Rationale The investigators are investigating the ability of near-infrared spectroscopy (NIRS) to detect altered brain function and oxygenation under a range of clinically relevant medical conditions.

NIRS allows for non-invasive measurement of oxygenated (O2Hb) and deoxygenated hemoglobin (HHb) concentrations in cortical brain tissue. Therefore, NIRS can be used to quantify cortical tissue oxygen saturation (StO2), which reflects changing metabolic rate and perfusion. Furthermore, functional NIRS (fNIRS) can be used to probe brain activity in a similar fashion to functional MRI, by assuming that the measured changes in blood perfusion and oxygenation are due to functional hyperemia (i.e. hemodynamic changes caused by neural activity). Using NIRS in patients, altered patterns of brain blood perfusion and reduced brain oxygenation levels have been shown to correlate with fatigue and impaired cognition, linking reduced cortical perfusion to symptoms that have been reported to occur in patients with IBD.

Tight regulation of cerebral blood flow is critical to ensure normal brain oxygenation and function. Cerebrovascular dysfunction and hypoxia have been implicated in a range of neurodegenerative and neuroinflammatory disorders including Alzheimer's disease and multiple sclerosis (MS). In a recent study using fNIRS, the investigators found altered task associated hemodynamic responses and brain hypoxia in patients with the immune-mediated liver disease, primary biliary cholangitis (PBC). Moreover, the experimental work in mice suggests that these changes may be due to the actions of TNFα on the cerebral vasculature. It also showed that patients with multiple sclerosis had reduced inter-hemispheric coherence and hypoxia. These observations led to the question of whether general systemic inflammation or brain/gut interactions could link to abnormal brain function and hypoxia, as detectable by NIRS.

Supporting this hypothesis is a recent NIRS study by Fujiwara T et al in patients with IBD. They showed that during performance of a task, mean oxygenated hemoglobin concentration was significantly lower in the frontal lobe in IBD patients compared to healthy controls. However, changes in brain oxygenation have not been previously examined during resting state or in the context of markers of peripheral inflammation, quality of life measures and symptom burden, or gut microbiome signatures in IBD patients.

This currently proposed substudy is to examine patients with inflammatory bowel disease (IBD) for their level of hypoxia, fNIRS functional response and fNIRS coherence.

IBD is increasing in incidence and prevalence worldwide. Several factors have been implicated in the development of IBD, including a dysregulated immune response to altered microbiota in a genetically susceptible host exposed to inciting environmental factors, but the specific cause of IBD remains unknown. Comorbid maladaptive behaviors and pain are prevalent in patients with IBD20-26. These mental health comorbidities complicate management of IBD, adversely impacting patient outcomes and health, and increasing the resource burden to the health care system. However, comorbid mental health issues and symptoms in IBD patients are poorly understood and under-treated, paralleling unmet mental health treatment needs in the general Canadian population. Therefore, an improved understanding of how brain changes occur in association with IBD, and their potential role in symptom development and link to systemic inflammation and gut microbiome signatures is of significant importance to improve management of these patients.

The gastrointestinal tract serves as a dynamic and local ecosystem for gut microbiota. Dysbiosis, which is an alteration of the gut microbial composition that contributes to host disease, occurs in IBD patients. Specifically, IBD patients exhibit a lower microbial α-diversity and are enriched in several groups of bacteria compared with healthy controls. Recently, preclinical, translational, and clinical studies have indicated that alterations in the structural composition or function of the microbiome can contribute to the development of mental illness, including depression-like behavior, and thus, is a vital component linking the gut-brain axis. Consistent with this, strong correlations have been identified between alterations in gut microbiota and the development of chronic inflammatory disorders, such as IBD, suggesting that dysbiosis is an important factor in both gastrointestinal disorders and mental health. However, the precise mechanisms by which gut dysbiosis in IBD may alter behavior remains poorly understood.

How peripheral inflammation, as occurs in IBD, leads to remote changes in brain function remains unclear and, as a result, there are limited therapeutic options available clinically to address this issue. A number of general pathways have been described that link systemic inflammation to changes occurring in the brain, which in turn give rise to altered behavior. These pathways traditionally have included signaling via neural pathways (mainly vagal nerve afferents) and immune signaling (mainly via circulating cytokines like TNFα, which either enter the brain directly or activate cerebral endothelium). Recently, University of Calgary researchers described a novel inflammation signaling pathway which involves increased peripheral TNF-α production driving increased microglial activation, followed by monocyte recruitment into brain vasculature and brain parenchyma, which in turn drives the development of sickness behaviors. TNFα is a multifunctional cytokine that mediates a range of effects that can directly impact brain function (via modulating neurotransmission) and the gut (e.g. affecting intestinal barrier permeability) and modulate tissue inflammation (e.g. activate macrophages to induce cytokine and chemokine expression). Increased circulating levels of TNFα and elevated production by circulating leukocytes are commonly documented in patients with chronic inflammatory conditions associated with a high prevalence of sickness behaviors and mood disorders, including IBD. Hence, blockade of TNFα signaling has been extensively evaluated in clinical studies of IBD. In addition, improvement in symptoms by TNFα signaling inhibition are often evident in treated patients with chronic inflammatory diseases, prior to overt changes in disease activity. In patients with IBD, anti-TNFα therapy was associated with significant improvements in sleep, depression, and anxiety early after initiation of therapy, and these improvements were sustained. Moreover, another study assessed the effect of anti-TNFα therapy on interoceptive signaling in patients with Crohn's disease and demonstrated reductions in visceral sensitivity and improved cognitive-affective processing after anti-TNFα administration, paralleled by improved sense of well being. Changes in cognition were linked to changes in neural activity in prefrontal and limbic brain areas. Moreover, the rapid behavioral and neural changes observed were not associated with significant changes in fecal calprotectin levels (marker of gut inflammation) suggesting they were unlikely related to a simultaneous reduction in intestinal inflammation. Anti-TNFα therapy also alters the gut microbiome in patients with IBD. Specifically, anti-TNFα therapy in IBD patients increased gut microbial species richness and phylodiversity to levels similar to healthy controls. In addition, anti-TNF therapy decreased the relative abundances of proinflammatory bacteria Escherichia and Enterococcus in IBD patients, and increasing genera that produce short-chain fatty acids, which have well-established anti-inflammatory effects in the gut.

Healthy cerebral endothelial cells (CECs) are critically important for brain blood flow regulation, as well as the normal function of the blood-brain barrier (BBB). Cytokines, including TNFα, originating from within the central nervous system or present in the peripheral blood circulation, can induce CEC dysfunction and increase BBB permeability, which is known to be associated with many neurological disorders including Alzheimer's and MS, as well as peripherally induced neuroinflammation. Indeed, CECs exposed to TNFα express fewer interendothelial proteins and have greater reactive oxygen species generation, leading to increased BBB permeability. Furthermore, CECs can be activated by cytokines that are either present in the blood or released by circulating immune cells in intimate contact with CECs, to produce secondary signaling molecules (e.g., additional cytokines, prostaglandin E2, nitric oxide) which interact with cells within the brain to alter NVC responses. Consistent with this suggestion, in a mouse model of peripheral inflammation, it was shown that activated monocytes within the cerebral circulation adhere to CECs and induce CEC activation through TNFα-TNF receptor-1 interactions. This immune cell and TNFα-driven CEC activation up-regulates inducible nitric oxide synthase expression within CECs and was directly linked to activation of microglia within the brain (especially those cells in close proximity to blood vessels), and ultimately to altered behavior. These previous findings from this group provide a mechanism by which peripheral inflammation can impact the function of CECs, thereby altering cerebrovascular function. Blocking activated immune cells within the circulation from adhering to CECs increases task-induced cortical blood flow (i.e., NVC)66, suggesting that immune cell-CEC adhesive interactions can lead to neurovascular uncoupling. CECs can also play an essential role in the regulation of cerebral blood flow by passively allowing vessel smooth muscle to relax and contract. Interestingly, activated leukocytes have been shown to promote endothelial cell-dependent vasospasticity and reduce arterial relaxation in vitro and in vivo. Further, endothelial cell-dependent vasospasticity is heightened in the presence of protein aggregates in the blood, which would effectively reduce the dynamic range of vasodilation. This is particularly interesting considering previous findings that peripheral inflammation leads to increased CEC presentation of the adhesion molecule P-selectin, which in turn promotes leukocyte and platelet adhesion to CECs. Taken together, these findings suggest that increased leukocyte-CEC interactions associated with peripheral inflammation may significantly contribute to altered cerebrovascular dynamics and potential neurovascular uncoupling in the setting of peripheral inflammatory disease, which is manifest as altered cerebral oxygenation.

Considered in the context of neuroinflammation associated with chronic peripheral inflammation, alterations in cortical perfusion and oxygenation may contribute, at least in part, to the behavioral symptoms associated with IBD and disease-associated reductions in health related quality of life (QoL).

The IBD clinic is routinely testing new treatments for IBD. They have agreed to integrate NIRS into a pilot protocol to determine if there is sufficient evidence to warrant a longer trial of NIRS as a biomarker of neurological involvement in IBD.

The investigators propose the following series of experiments, using NIRS, to determine (A) whether patients with IBD exhibit reduced cortical oxygen saturation and altered patterns of microvascular cerebral blood perfusion; (B) whether NIRS findings of oxygen saturation and perfusion correlate with clinical disease activity markers, a disease-specific gut microbiome signature, and/or symptom and quality of life scores in patients with IBD; (C) the impact of anti-TNF therapy (administered as clinically indicated, as standard of practice) on NIRS changes, the fecal microbiome, markers of systemic inflammation, and symptom severity.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will be:

* > 18 years of age with moderate-to-severe UC or (partial Mayo score [excluding endoscopy] ≥5 with rectal bleeding subscore ≥1; or total Mayo subscore 6-12 with RBS ≥1) or CD (Harvey-Bradshaw index [HBI] of 7 or greater, and active CD confirmed on POC bowel ultrasound (defined by bowel wall thickness >3mm and positive Color doppler signal and a fecal calprotectin > 50 μg/g ).
* based on their active disease status patients cannot be taking > 20 mg prednisone daily and
* must be eligible for anti-TNF therapy as per standard of care (clinical decision made by IBD specialist caring for the patient).

Exclusion Criteria:

* patients with severely active UC (clinical signs of fulminant colitis or toxic megacolon) or CD (HBI > 16), requiring > 20 mg of prednisone daily at induction, suicidal ideation or psychosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have either Ulcerative Colitis or Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-26 (Estimated); Primary Completion 2025-01-05 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
a) Clinically: CD (decrease of >3 points in the modified Harvey-Bradshaw Index); UC (decrease of >2 points in the partial Mayo Score) | 16 weeks
  Defining differences in alterations of resting state brain NIRS findings occurring in IBD patients, between baseline and at 16 weeks after starting anti-TNF therapy, in anti-TNF responders vs. non-responders, defined:
  a) Clinically: CD (decrease of >3 points in the modified Harvey-Bradshaw Index); UC (decrease of >2 points in the partial Mayo Score)
b) Radiographically: decrease in bowel wall thickness ≥25% in most affected segment with 2 point decrease in color Doppler signal score or normalization | 16 weeks
  Defining differences in alterations of resting state brain NIRS findings occurring in IBD patients, between baseline and at 16 weeks after starting anti-TNF therapy, in anti-TNF responders vs. non-responders, defined:
  b) Radiographically: decrease in bowel wall thickness ≥25% in most affected segment with 2 point decrease in color Doppler signal score or normalization
c) Biomarker: decrease in fecal calprotectin >50% from baseline or ≤250 ug/g | 16 weeks
  Defining differences in alterations of resting state brain NIRS findings occurring in IBD patients, between baseline and at 16 weeks after starting anti-TNF therapy, in anti-TNF responders vs. non-responders, defined:
  c) Biomarker: decrease in fecal calprotectin >50% from baseline or ≤250 ug/g
d) Endoscopically (where available): CD (decrease in Simple Endoscopic Score for CD ≥50% from baseline); UC (decrease in Mayo endoscopic subscore ≥1 point from baseline) | 16 weeks
  Defining differences in alterations of resting state brain NIRS findings occurring in IBD patients, between baseline and at 16 weeks after starting anti-TNF therapy, in anti-TNF responders vs. non-responders, defined:
  d) Endoscopically (where available): CD (decrease in Simple Endoscopic Score for CD ≥50% from baseline); UC (decrease in Mayo endoscopic subscore ≥1 point from baseline)

SECONDARY OUTCOMES:
(i) alterations in markers of bowel (defined by bowel ultrasound) and systemic inflammation. | 16 weeks
  Delineating whether baseline brain NIRS findings, and changes in NIRS findings from baseline to 16 weeks after starting anti-TNF therapy, correlate with:
  (i) alterations in markers of bowel (defined by bowel ultrasound) and systemic inflammation.
(ii) reduction from baseline measurement of fecal calprotectin level. | 16 weeks
  Delineating whether baseline brain NIRS findings, and changes in NIRS findings from baseline to 16 weeks after starting anti-TNF therapy, correlate with:
  (ii) reduction from baseline measurement of fecal calprotectin level.
(iii) specific gut microbiome and metabolomics signatures. | 16 weeks
  Delineating whether baseline brain NIRS findings, and changes in NIRS findings from baseline to 16 weeks after starting anti-TNF therapy, correlate with:
  (iii) specific gut microbiome and metabolomics signatures.
(iv) changes in symptom severity in IBD patients that respond (defined as above), or do not respond to anti-TNF therapy. | 16 weeks
  Delineating whether baseline brain NIRS findings, and changes in NIRS findings from baseline to 16 weeks after starting anti-TNF therapy, correlate with:
  (iv) changes in symptom severity in IBD patients that respond (defined as above), or do not respond to anti-TNF therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Swain, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scholkmann F, Kleiser S, Metz AJ, Zimmermann R, Mata Pavia J, Wolf U, Wolf M. A review on continuous wave functional near-infrared spectroscopy and imaging instrumentation and methodology. Neuroimage. 2014 Jan 15;85 Pt 1:6-27. doi: 10.1016/j.neuroimage.2013.05.004. Epub 2013 May 16. PMID 23684868
- [Background] Sokoloff L. Local cerebral energy metabolism: its relationships to local functional activity and blood flow. Ciba Found Symp. 1978 Mar;(56):171-97. doi: 10.1002/9780470720370.ch10. PMID 97062
- [Background] Nippert AR, Biesecker KR, Newman EA. Mechanisms Mediating Functional Hyperemia in the Brain. Neuroscientist. 2018 Feb;24(1):73-83. doi: 10.1177/1073858417703033. Epub 2017 Apr 12. PMID 28403673
- [Background] Nippert AR, Mishra A, Newman EA. Keeping the Brain Well Fed: The Role of Capillaries and Arterioles in Orchestrating Functional Hyperemia. Neuron. 2018 Jul 25;99(2):248-250. doi: 10.1016/j.neuron.2018.07.011. PMID 30048612
- [Background] Bu L, Zhang M, Li J, Li F, Liu H, Li Z. Effects of Sleep Deprivation on Phase Synchronization as Assessed by Wavelet Phase Coherence Analysis of Prefrontal Tissue Oxyhemoglobin Signals. PLoS One. 2017 Jan 3;12(1):e0169279. doi: 10.1371/journal.pone.0169279. eCollection 2017. PMID 28046043
- [Background] Tarumi T, Dunsky DI, Khan MA, Liu J, Hill C, Armstrong K, Martin-Cook K, Cullum CM, Zhang R. Dynamic cerebral autoregulation and tissue oxygenation in amnestic mild cognitive impairment. J Alzheimers Dis. 2014;41(3):765-78. doi: 10.3233/JAD-132018. PMID 24670396
- [Background] Uemura K, Shimada H, Doi T, Makizako H, Tsutsumimoto K, Park H, Suzuki T. Reduced prefrontal oxygenation in mild cognitive impairment during memory retrieval. Int J Geriatr Psychiatry. 2016 Jun;31(6):583-91. doi: 10.1002/gps.4363. Epub 2015 Sep 21. PMID 26387497
- [Background] Shang J, Yamashita T, Zhai Y, Nakano Y, Morihara R, Fukui Y, Hishikawa N, Ohta Y, Abe K. Strong Impact of Chronic Cerebral Hypoperfusion on Neurovascular Unit, Cerebrovascular Remodeling, and Neurovascular Trophic Coupling in Alzheimer's Disease Model Mouse. J Alzheimers Dis. 2016 Mar 5;52(1):113-26. doi: 10.3233/JAD-151126. PMID 27060955
- [Background] Yang R, Dunn JF. Reduced cortical microvascular oxygenation in multiple sclerosis: a blinded, case-controlled study using a novel quantitative near-infrared spectroscopy method. Sci Rep. 2015 Nov 13;5:16477. doi: 10.1038/srep16477. PMID 26563581
- [Background] Duszynski CC, Avati V, Lapointe AP, Scholkmann F, Dunn JF, Swain MG. Near-Infrared Spectroscopy Reveals Brain Hypoxia and Cerebrovascular Dysregulation in Primary Biliary Cholangitis. Hepatology. 2020 Apr;71(4):1408-1420. doi: 10.1002/hep.30920. Epub 2019 Dec 31. PMID 31535726
- [Background] D'Mello C, Le T, Swain MG. Cerebral microglia recruit monocytes into the brain in response to tumor necrosis factoralpha signaling during peripheral organ inflammation. J Neurosci. 2009 Feb 18;29(7):2089-102. doi: 10.1523/JNEUROSCI.3567-08.2009. PMID 19228962
- [Background] Fujiwara T, Kono S, Katakura K, Abe K, Takahashi A, Gunji N, Yokokawa A, Kawashima K, Suzuki R, Wada A, Miura I, Yabe H, Ohira H. Evaluation of Brain Activity Using Near-infrared Spectroscopy in Inflammatory Bowel Disease Patients. Sci Rep. 2018 Jan 10;8(1):402. doi: 10.1038/s41598-017-18897-4. PMID 29321655
- [Background] Kaplan GG. The global burden of IBD: from 2015 to 2025. Nat Rev Gastroenterol Hepatol. 2015 Dec;12(12):720-7. doi: 10.1038/nrgastro.2015.150. Epub 2015 Sep 1. PMID 26323879
- [Background] Kaplan GG, Bernstein CN, Coward S, Bitton A, Murthy SK, Nguyen GC, Lee K, Cooke-Lauder J, Benchimol EI. The Impact of Inflammatory Bowel Disease in Canada 2018: Epidemiology. J Can Assoc Gastroenterol. 2019 Feb;2(Suppl 1):S6-S16. doi: 10.1093/jcag/gwy054. Epub 2018 Nov 2. PMID 31294381
- [Background] Khor B, Gardet A, Xavier RJ. Genetics and pathogenesis of inflammatory bowel disease. Nature. 2011 Jun 15;474(7351):307-17. doi: 10.1038/nature10209. PMID 21677747
- [Background] Halfvarson J, Brislawn CJ, Lamendella R, Vazquez-Baeza Y, Walters WA, Bramer LM, D'Amato M, Bonfiglio F, McDonald D, Gonzalez A, McClure EE, Dunklebarger MF, Knight R, Jansson JK. Dynamics of the human gut microbiome in inflammatory bowel disease. Nat Microbiol. 2017 Feb 13;2:17004. doi: 10.1038/nmicrobiol.2017.4. PMID 28191884
- [Background] Ni J, Wu GD, Albenberg L, Tomov VT. Gut microbiota and IBD: causation or correlation? Nat Rev Gastroenterol Hepatol. 2017 Oct;14(10):573-584. doi: 10.1038/nrgastro.2017.88. Epub 2017 Jul 19. PMID 28743984
- [Background] Lavelle A, Sokol H. Gut microbiota: Beyond metagenomics, metatranscriptomics illuminates microbiome functionality in IBD. Nat Rev Gastroenterol Hepatol. 2018 Apr;15(4):193-194. doi: 10.1038/nrgastro.2018.15. Epub 2018 Feb 21. No abstract available. PMID 29463904
- [Background] Knights D, Lassen KG, Xavier RJ. Advances in inflammatory bowel disease pathogenesis: linking host genetics and the microbiome. Gut. 2013 Oct;62(10):1505-10. doi: 10.1136/gutjnl-2012-303954. PMID 24037875
- [Background] Moradkhani A, Beckman LJ, Tabibian JH. Health-related quality of life in inflammatory bowel disease: psychosocial, clinical, socioeconomic, and demographic predictors. J Crohns Colitis. 2013 Jul;7(6):467-73. doi: 10.1016/j.crohns.2012.07.012. Epub 2012 Aug 10. PMID 22884758
- [Background] Nocerino A, Nguyen A, Agrawal M, Mone A, Lakhani K, Swaminath A. Fatigue in Inflammatory Bowel Diseases: Etiologies and Management. Adv Ther. 2020 Jan;37(1):97-112. doi: 10.1007/s12325-019-01151-w. Epub 2019 Nov 23. PMID 31760611
- [Background] Graff LA, Walker JR, Lix L, Clara I, Rawsthorne P, Rogala L, Miller N, Jakul L, McPhail C, Ediger J, Bernstein CN. The relationship of inflammatory bowel disease type and activity to psychological functioning and quality of life. Clin Gastroenterol Hepatol. 2006 Dec;4(12):1491-1501. doi: 10.1016/j.cgh.2006.09.027. PMID 17162241
- [Background] Bonaz BL, Bernstein CN. Brain-gut interactions in inflammatory bowel disease. Gastroenterology. 2013 Jan;144(1):36-49. doi: 10.1053/j.gastro.2012.10.003. Epub 2012 Oct 12. PMID 23063970
- [Background] Szigethy E. Pain Management in Patients With Inflammatory Bowel Disease. Gastroenterol Hepatol (N Y). 2018 Jan;14(1):53-56. No abstract available. PMID 29491764
- [Background] Hashash JG, Ramos-Rivers C, Youk A, Chiu WK, Duff K, Regueiro M, Binion DG, Koutroubakis I, Vachon A, Benhayon D, Dunn MA, Szigethy EM. Quality of Sleep and Coexistent Psychopathology Have Significant Impact on Fatigue Burden in Patients With Inflammatory Bowel Disease. J Clin Gastroenterol. 2018 May/Jun;52(5):423-430. doi: 10.1097/MCG.0000000000000729. PMID 27775960
- [Background] Jones JL, Nguyen GC, Benchimol EI, Bernstein CN, Bitton A, Kaplan GG, Murthy SK, Lee K, Cooke-Lauder J, Otley AR. The Impact of Inflammatory Bowel Disease in Canada 2018: Quality of Life. J Can Assoc Gastroenterol. 2019 Feb;2(Suppl 1):S42-S48. doi: 10.1093/jcag/gwy048. Epub 2018 Nov 2. PMID 31294384
- [Background] Kuenzig ME, Benchimol EI, Lee L, Targownik LE, Singh H, Kaplan GG, Bernstein CN, Bitton A, Nguyen GC, Lee K, Cooke-Lauder J, Murthy SK. The Impact of Inflammatory Bowel Disease in Canada 2018: Direct Costs and Health Services Utilization. J Can Assoc Gastroenterol. 2019 Feb;2(Suppl 1):S17-S33. doi: 10.1093/jcag/gwy055. Epub 2018 Nov 2. PMID 31294382
- [Background] Kuenzig ME, Lee L, El-Matary W, Weizman AV, Benchimol EI, Kaplan GG, Nguyen GC, Bernstein CN, Bitton A, Lee K, Cooke-Lauder J, Murthy SK. The Impact of Inflammatory Bowel Disease in Canada 2018: Indirect Costs of IBD Care. J Can Assoc Gastroenterol. 2019 Feb;2(Suppl 1):S34-S41. doi: 10.1093/jcag/gwy050. Epub 2018 Nov 2. PMID 31294383
- [Background] Cryan JF, O'Riordan KJ, Cowan CSM, Sandhu KV, Bastiaanssen TFS, Boehme M, Codagnone MG, Cussotto S, Fulling C, Golubeva AV, Guzzetta KE, Jaggar M, Long-Smith CM, Lyte JM, Martin JA, Molinero-Perez A, Moloney G, Morelli E, Morillas E, O'Connor R, Cruz-Pereira JS, Peterson VL, Rea K, Ritz NL, Sherwin E, Spichak S, Teichman EM, van de Wouw M, Ventura-Silva AP, Wallace-Fitzsimons SE, Hyland N, Clarke G, Dinan TG. The Microbiota-Gut-Brain Axis. Physiol Rev. 2019 Oct 1;99(4):1877-2013. doi: 10.1152/physrev.00018.2018. PMID 31460832
- [Background] Somineni HK, Kugathasan S. The Microbiome in Patients With Inflammatory Diseases. Clin Gastroenterol Hepatol. 2019 Jan;17(2):243-255. doi: 10.1016/j.cgh.2018.08.078. Epub 2018 Sep 7. PMID 30196163
- [Background] Ott SJ, Musfeldt M, Wenderoth DF, Hampe J, Brant O, Folsch UR, Timmis KN, Schreiber S. Reduction in diversity of the colonic mucosa associated bacterial microflora in patients with active inflammatory bowel disease. Gut. 2004 May;53(5):685-93. doi: 10.1136/gut.2003.025403. PMID 15082587
- [Background] Pascal V, Pozuelo M, Borruel N, Casellas F, Campos D, Santiago A, Martinez X, Varela E, Sarrabayrouse G, Machiels K, Vermeire S, Sokol H, Guarner F, Manichanh C. A microbial signature for Crohn's disease. Gut. 2017 May;66(5):813-822. doi: 10.1136/gutjnl-2016-313235. Epub 2017 Feb 7. PMID 28179361
- [Background] Guida F, Turco F, Iannotta M, De Gregorio D, Palumbo I, Sarnelli G, Furiano A, Napolitano F, Boccella S, Luongo L, Mazzitelli M, Usiello A, De Filippis F, Iannotti FA, Piscitelli F, Ercolini D, de Novellis V, Di Marzo V, Cuomo R, Maione S. Antibiotic-induced microbiota perturbation causes gut endocannabinoidome changes, hippocampal neuroglial reorganization and depression in mice. Brain Behav Immun. 2018 Jan;67:230-245. doi: 10.1016/j.bbi.2017.09.001. Epub 2017 Sep 7. PMID 28890155
- [Background] Zheng P, Zeng B, Zhou C, Liu M, Fang Z, Xu X, Zeng L, Chen J, Fan S, Du X, Zhang X, Yang D, Yang Y, Meng H, Li W, Melgiri ND, Licinio J, Wei H, Xie P. Gut microbiome remodeling induces depressive-like behaviors through a pathway mediated by the host's metabolism. Mol Psychiatry. 2016 Jun;21(6):786-96. doi: 10.1038/mp.2016.44. Epub 2016 Apr 12. PMID 27067014
- [Background] Mi GL, Zhao L, Qiao DD, Kang WQ, Tang MQ, Xu JK. Effectiveness of Lactobacillus reuteri in infantile colic and colicky induced maternal depression: a prospective single blind randomized trial. Antonie Van Leeuwenhoek. 2015 Jun;107(6):1547-53. doi: 10.1007/s10482-015-0448-9. Epub 2015 Apr 16. PMID 25876529
- [Background] Cryan JF, Dinan TG. Mind-altering microorganisms: the impact of the gut microbiota on brain and behaviour. Nat Rev Neurosci. 2012 Oct;13(10):701-12. doi: 10.1038/nrn3346. Epub 2012 Sep 12. PMID 22968153
- [Background] Bravo JA, Julio-Pieper M, Forsythe P, Kunze W, Dinan TG, Bienenstock J, Cryan JF. Communication between gastrointestinal bacteria and the nervous system. Curr Opin Pharmacol. 2012 Dec;12(6):667-72. doi: 10.1016/j.coph.2012.09.010. Epub 2012 Oct 4. PMID 23041079
- [Background] Zhang M, Sun K, Wu Y, Yang Y, Tso P, Wu Z. Interactions between Intestinal Microbiota and Host Immune Response in Inflammatory Bowel Disease. Front Immunol. 2017 Aug 14;8:942. doi: 10.3389/fimmu.2017.00942. eCollection 2017. PMID 28855901
- [Background] Collins SM. Interrogating the Gut-Brain Axis in the Context of Inflammatory Bowel Disease: A Translational Approach. Inflamm Bowel Dis. 2020 Mar 4;26(4):493-501. doi: 10.1093/ibd/izaa004. PMID 31970390
- [Background] Thomann AK, Mak JWY, Zhang JW, Wuestenberg T, Ebert MP, Sung JJY, Bernstein CN, Reindl W, Ng SC. Review article: bugs, inflammation and mood-a microbiota-based approach to psychiatric symptoms in inflammatory bowel diseases. Aliment Pharmacol Ther. 2020 Jul;52(2):247-266. doi: 10.1111/apt.15787. Epub 2020 Jun 11. PMID 32525605
- [Background] Capuron L, Miller AH. Immune system to brain signaling: neuropsychopharmacological implications. Pharmacol Ther. 2011 May;130(2):226-38. doi: 10.1016/j.pharmthera.2011.01.014. Epub 2011 Feb 17. PMID 21334376
- [Background] D'Mello C, Swain MG. Liver-brain interactions in inflammatory liver diseases: implications for fatigue and mood disorders. Brain Behav Immun. 2014 Jan;35:9-20. doi: 10.1016/j.bbi.2013.10.009. Epub 2013 Oct 16. PMID 24140301
- [Background] D'Mello C, Swain MG. Immune-to-Brain Communication Pathways in Inflammation-Associated Sickness and Depression. Curr Top Behav Neurosci. 2017;31:73-94. doi: 10.1007/7854_2016_37. PMID 27677781
- [Background] D'Mello C, Riazi K, Le T, Stevens KM, Wang A, McKay DM, Pittman QJ, Swain MG. P-selectin-mediated monocyte-cerebral endothelium adhesive interactions link peripheral organ inflammation to sickness behaviors. J Neurosci. 2013 Sep 11;33(37):14878-88. doi: 10.1523/JNEUROSCI.1329-13.2013. PMID 24027287
- [Background] Chu WM. Tumor necrosis factor. Cancer Lett. 2013 Jan 28;328(2):222-5. doi: 10.1016/j.canlet.2012.10.014. Epub 2012 Oct 22. PMID 23085193
- [Background] Sedger LM, McDermott MF. TNF and TNF-receptors: From mediators of cell death and inflammation to therapeutic giants - past, present and future. Cytokine Growth Factor Rev. 2014 Aug;25(4):453-72. doi: 10.1016/j.cytogfr.2014.07.016. Epub 2014 Aug 1. PMID 25169849
- [Background] Padmos RC, Hillegers MH, Knijff EM, Vonk R, Bouvy A, Staal FJ, de Ridder D, Kupka RW, Nolen WA, Drexhage HA. A discriminating messenger RNA signature for bipolar disorder formed by an aberrant expression of inflammatory genes in monocytes. Arch Gen Psychiatry. 2008 Apr;65(4):395-407. doi: 10.1001/archpsyc.65.4.395. PMID 18391128
- [Background] Slebioda TJ, Kmiec Z. Tumour necrosis factor superfamily members in the pathogenesis of inflammatory bowel disease. Mediators Inflamm. 2014;2014:325129. doi: 10.1155/2014/325129. Epub 2014 Jun 17. PMID 25045210
- [Background] Singh UP, Singh NP, Murphy EA, Price RL, Fayad R, Nagarkatti M, Nagarkatti PS. Chemokine and cytokine levels in inflammatory bowel disease patients. Cytokine. 2016 Jan;77:44-9. doi: 10.1016/j.cyto.2015.10.008. Epub 2015 Oct 29. PMID 26520877
- [Background] Muzes G, Molnar B, Tulassay Z, Sipos F. Changes of the cytokine profile in inflammatory bowel diseases. World J Gastroenterol. 2012 Nov 7;18(41):5848-61. doi: 10.3748/wjg.v18.i41.5848. PMID 23139600
- [Background] Lichtenstein GR. Comprehensive review: antitumor necrosis factor agents in inflammatory bowel disease and factors implicated in treatment response. Therap Adv Gastroenterol. 2013 Jul;6(4):269-93. doi: 10.1177/1756283X13479826. PMID 23814608
- [Background] Gray MA, Chao CY, Staudacher HM, Kolosky NA, Talley NJ, Holtmann G. Anti-TNFalpha therapy in IBD alters brain activity reflecting visceral sensory function and cognitive-affective biases. PLoS One. 2018 Mar 8;13(3):e0193542. doi: 10.1371/journal.pone.0193542. eCollection 2018. PMID 29518097
- [Background] Lichtenstein GR, Bala M, Han C, DeWoody K, Schaible T. Infliximab improves quality of life in patients with Crohn's disease. Inflamm Bowel Dis. 2002 Jul;8(4):237-43. doi: 10.1097/00054725-200207000-00001. PMID 12131606
- [Background] Horst S, Chao A, Rosen M, Nohl A, Duley C, Wagnon JH, Beaulieu DB, Taylor W, Gaines L, Schwartz DA. Treatment with immunosuppressive therapy may improve depressive symptoms in patients with inflammatory bowel disease. Dig Dis Sci. 2015 Feb;60(2):465-70. doi: 10.1007/s10620-014-3375-0. Epub 2014 Oct 2. PMID 25274158
- [Background] Stevens BW, Borren NZ, Velonias G, Conway G, Cleland T, Andrews E, Khalili H, Garber JG, Xavier RJ, Yajnik V, Ananthakrishnan AN. Vedolizumab Therapy Is Associated with an Improvement in Sleep Quality and Mood in Inflammatory Bowel Diseases. Dig Dis Sci. 2017 Jan;62(1):197-206. doi: 10.1007/s10620-016-4356-2. Epub 2016 Oct 28. PMID 27796768
- [Background] Wang F, Lin X, Zhao Q, Li J. Adverse symptoms with anti-TNF-alpha therapy in inflammatory bowel disease: systematic review and duration-response meta-analysis. Eur J Clin Pharmacol. 2015 Aug;71(8):911-9. doi: 10.1007/s00228-015-1877-0. Epub 2015 May 30. PMID 26022220
- [Background] Aden K, Rehman A, Waschina S, Pan WH, Walker A, Lucio M, Nunez AM, Bharti R, Zimmerman J, Bethge J, Schulte B, Schulte D, Franke A, Nikolaus S, Schroeder JO, Vandeputte D, Raes J, Szymczak S, Waetzig GH, Zeuner R, Schmitt-Kopplin P, Kaleta C, Schreiber S, Rosenstiel P. Metabolic Functions of Gut Microbes Associate With Efficacy of Tumor Necrosis Factor Antagonists in Patients With Inflammatory Bowel Diseases. Gastroenterology. 2019 Nov;157(5):1279-1292.e11. doi: 10.1053/j.gastro.2019.07.025. Epub 2019 Jul 18. PMID 31326413
- [Background] Estevinho MM, Rocha C, Correia L, Lago P, Ministro P, Portela F, Trindade E, Afonso J, Peyrin-Biroulet L, Magro F; GEDII (Portuguese IBD Group). Features of Fecal and Colon Microbiomes Associate With Responses to Biologic Therapies for Inflammatory Bowel Diseases: A Systematic Review. Clin Gastroenterol Hepatol. 2020 May;18(5):1054-1069. doi: 10.1016/j.cgh.2019.08.063. Epub 2019 Sep 14. PMID 31526845
- [Background] Kisler K, Nelson AR, Montagne A, Zlokovic BV. Cerebral blood flow regulation and neurovascular dysfunction in Alzheimer disease. Nat Rev Neurosci. 2017 Jul;18(7):419-434. doi: 10.1038/nrn.2017.48. Epub 2017 May 18. PMID 28515434
- [Background] Correale J, Villa A. The blood-brain-barrier in multiple sclerosis: functional roles and therapeutic targeting. Autoimmunity. 2007 Mar;40(2):148-60. doi: 10.1080/08916930601183522. PMID 17453713
- [Background] Rochfort KD, Collins LE, Murphy RP, Cummins PM. Downregulation of blood-brain barrier phenotype by proinflammatory cytokines involves NADPH oxidase-dependent ROS generation: consequences for interendothelial adherens and tight junctions. PLoS One. 2014 Jul 3;9(7):e101815. doi: 10.1371/journal.pone.0101815. eCollection 2014. PMID 24992685
- [Background] Akopov S, Sercombe R, Seylaz J. Cerebrovascular reactivity: role of endothelium/platelet/leukocyte interactions. Cerebrovasc Brain Metab Rev. 1996 Spring;8(1):11-94. PMID 9052980
- [Background] Tohidpour A, Morgun AV, Boitsova EB, Malinovskaya NA, Martynova GP, Khilazheva ED, Kopylevich NV, Gertsog GE, Salmina AB. Neuroinflammation and Infection: Molecular Mechanisms Associated with Dysfunction of Neurovascular Unit. Front Cell Infect Microbiol. 2017 Jun 20;7:276. doi: 10.3389/fcimb.2017.00276. eCollection 2017. PMID 28676848
- [Background] Kerfoot SM, D'Mello C, Nguyen H, Ajuebor MN, Kubes P, Le T, Swain MG. TNF-alpha-secreting monocytes are recruited into the brain of cholestatic mice. Hepatology. 2006 Jan;43(1):154-62. doi: 10.1002/hep.21003. PMID 16374849
- [Background] D'Mello C, Almishri W, Liu H, Swain MG. Interactions Between Platelets and Inflammatory Monocytes Affect Sickness Behavior in Mice With Liver Inflammation. Gastroenterology. 2017 Nov;153(5):1416-1428.e2. doi: 10.1053/j.gastro.2017.08.011. Epub 2017 Aug 9. PMID 28802564
- [Background] Reinhard M, Rosengarten B, Kirchhoff L, Hetzel A, Rauer S. Natalizumab and regulation of cerebral blood flow: results from an observational study. Eur Neurol. 2010;64(2):124-8. doi: 10.1159/000316765. Epub 2010 Jul 22. PMID 20664205
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Moskovitz DN, Daperno M, Van Assche GA, et al. Defining and validating cut-offs for the simple endoscopic score for Crohn's disease. Gastroenterology 2007;132:A173-A173.
- [Background] Limberg B. [Diagnosis of chronic inflammatory bowel disease by ultrasonography]. Z Gastroenterol. 1999 Jun;37(6):495-508. German. PMID 10427656
- [Background] Walsham NE, Sherwood RA. Fecal calprotectin in inflammatory bowel disease. Clin Exp Gastroenterol. 2016 Jan 28;9:21-9. doi: 10.2147/CEG.S51902. eCollection 2016. PMID 26869808
- [Background] Walmsley RS, Ayres RC, Pounder RE, Allan RN. A simple clinical colitis activity index. Gut. 1998 Jul;43(1):29-32. doi: 10.1136/gut.43.1.29. PMID 9771402
- [Background] Harvey RF, Bradshaw JM. A simple index of Crohn's-disease activity. Lancet. 1980 Mar 8;1(8167):514. doi: 10.1016/s0140-6736(80)92767-1. No abstract available. PMID 6102236
- [Background] Irvine EJ, Zhou Q, Thompson AK. The Short Inflammatory Bowel Disease Questionnaire: a quality of life instrument for community physicians managing inflammatory bowel disease. CCRPT Investigators. Canadian Crohn's Relapse Prevention Trial. Am J Gastroenterol. 1996 Aug;91(8):1571-8. PMID 8759664
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spiegel BM, Hays RD, Bolus R, Melmed GY, Chang L, Whitman C, Khanna PP, Paz SH, Hays T, Reise S, Khanna D. Development of the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) gastrointestinal symptom scales. Am J Gastroenterol. 2014 Nov;109(11):1804-14. doi: 10.1038/ajg.2014.237. Epub 2014 Sep 9. PMID 25199473
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Osman A, Barrios FX, Gutierrez PM, Kopper BA, Merrifield T, Grittmann L. The Pain Catastrophizing Scale: further psychometric evaluation with adult samples. J Behav Med. 2000 Aug;23(4):351-65. doi: 10.1023/a:1005548801037. PMID 10984864
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] van Tilburg Bernardes E, Pettersen VK, Gutierrez MW, Laforest-Lapointe I, Jendzjowsky NG, Cavin JB, Vicentini FA, Keenan CM, Ramay HR, Samara J, MacNaughton WK, Wilson RJA, Kelly MM, McCoy KD, Sharkey KA, Arrieta MC. Intestinal fungi are causally implicated in microbiome assembly and immune development in mice. Nat Commun. 2020 May 22;11(1):2577. doi: 10.1038/s41467-020-16431-1. PMID 32444671
- [Background] Arrieta MC, Arevalo A, Stiemsma L, Dimitriu P, Chico ME, Loor S, Vaca M, Boutin RCT, Morien E, Jin M, Turvey SE, Walter J, Parfrey LW, Cooper PJ, Finlay B. Associations between infant fungal and bacterial dysbiosis and childhood atopic wheeze in a nonindustrialized setting. J Allergy Clin Immunol. 2018 Aug;142(2):424-434.e10. doi: 10.1016/j.jaci.2017.08.041. Epub 2017 Dec 11. PMID 29241587
- [Background] Tan Q, Zhang M, Wang Y, Zhang M, Wang Y, Xin Q, Wang B, Li Z. Frequency-specific functional connectivity revealed by wavelet-based coherence analysis in elderly subjects with cerebral infarction using NIRS method. Med Phys. 2015 Sep;42(9):5391-403. doi: 10.1118/1.4928672. PMID 26328988
- [Background] Chang C, Glover GH. Time-frequency dynamics of resting-state brain connectivity measured with fMRI. Neuroimage. 2010 Mar;50(1):81-98. doi: 10.1016/j.neuroimage.2009.12.011. Epub 2009 Dec 16. PMID 20006716
- [Background] Julien C. The enigma of Mayer waves: Facts and models. Cardiovasc Res. 2006 Apr 1;70(1):12-21. doi: 10.1016/j.cardiores.2005.11.008. Epub 2005 Dec 19. PMID 16360130
- [Background] Fox MD, Raichle ME. Spontaneous fluctuations in brain activity observed with functional magnetic resonance imaging. Nat Rev Neurosci. 2007 Sep;8(9):700-11. doi: 10.1038/nrn2201. PMID 17704812
- [Background] Birn RM, Diamond JB, Smith MA, Bandettini PA. Separating respiratory-variation-related fluctuations from neuronal-activity-related fluctuations in fMRI. Neuroimage. 2006 Jul 15;31(4):1536-48. doi: 10.1016/j.neuroimage.2006.02.048. Epub 2006 Apr 24. PMID 16632379
- [Background] Wise RG, Ide K, Poulin MJ, Tracey I. Resting fluctuations in arterial carbon dioxide induce significant low frequency variations in BOLD signal. Neuroimage. 2004 Apr;21(4):1652-64. doi: 10.1016/j.neuroimage.2003.11.025. PMID 15050588
- [Background] Gatto R, Hoffman W, Mueller M, Flores A, Valyi-Nagy T, Charbel FT. Frequency domain near-infrared spectroscopy technique in the assessment of brain oxygenation: a validation study in live subjects and cadavers. J Neurosci Methods. 2006 Oct 30;157(2):274-7. doi: 10.1016/j.jneumeth.2006.04.013. Epub 2006 May 24. PMID 16730069
- [Background] Novak KL, Kaplan GG, Panaccione R, Afshar EE, Tanyingoh D, Swain M, Kellar A, Wilson S. A Simple Ultrasound Score for the Accurate Detection of Inflammatory Activity in Crohn's Disease. Inflamm Bowel Dis. 2017 Nov;23(11):2001-2010. doi: 10.1097/MIB.0000000000001174. PMID 28644185
- [Background] WILCOXON F. Individual comparisons of grouped data by ranking methods. J Econ Entomol. 1946 Apr;39:269. doi: 10.1093/jee/39.2.269. No abstract available. PMID 20983181
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Bartram AK, Lynch MD, Stearns JC, Moreno-Hagelsieb G, Neufeld JD. Generation of multimillion-sequence 16S rRNA gene libraries from complex microbial communities by assembling paired-end illumina reads. Appl Environ Microbiol. 2011 Jun;77(11):3846-52. doi: 10.1128/AEM.02772-10. Epub 2011 Apr 1. PMID 21460107
- [Background] Schloss PD, Westcott SL, Ryabin T, Hall JR, Hartmann M, Hollister EB, Lesniewski RA, Oakley BB, Parks DH, Robinson CJ, Sahl JW, Stres B, Thallinger GG, Van Horn DJ, Weber CF. Introducing mothur: open-source, platform-independent, community-supported software for describing and comparing microbial communities. Appl Environ Microbiol. 2009 Dec;75(23):7537-41. doi: 10.1128/AEM.01541-09. Epub 2009 Oct 2. PMID 19801464
- [Background] DeSantis TZ, Hugenholtz P, Larsen N, Rojas M, Brodie EL, Keller K, Huber T, Dalevi D, Hu P, Andersen GL. Greengenes, a chimera-checked 16S rRNA gene database and workbench compatible with ARB. Appl Environ Microbiol. 2006 Jul;72(7):5069-72. doi: 10.1128/AEM.03006-05. PMID 16820507
- [Background] McMurdie PJ, Holmes S. phyloseq: an R package for reproducible interactive analysis and graphics of microbiome census data. PLoS One. 2013 Apr 22;8(4):e61217. doi: 10.1371/journal.pone.0061217. Print 2013. PMID 23630581
- [Background] McMurdie PJ, Holmes S. Waste not, want not: why rarefying microbiome data is inadmissible. PLoS Comput Biol. 2014 Apr 3;10(4):e1003531. doi: 10.1371/journal.pcbi.1003531. eCollection 2014 Apr. PMID 24699258
- [Background] Love MI, Huber W, Anders S. Moderated estimation of fold change and dispersion for RNA-seq data with DESeq2. Genome Biol. 2014;15(12):550. doi: 10.1186/s13059-014-0550-8. PMID 25516281
- [Background] Morgan XC, Tickle TL, Sokol H, Gevers D, Devaney KL, Ward DV, Reyes JA, Shah SA, LeLeiko N, Snapper SB, Bousvaros A, Korzenik J, Sands BE, Xavier RJ, Huttenhower C. Dysfunction of the intestinal microbiome in inflammatory bowel disease and treatment. Genome Biol. 2012 Apr 16;13(9):R79. doi: 10.1186/gb-2012-13-9-r79. PMID 23013615
- [Background] B Sohn M, Li H. A GLM-based latent variable ordination method for microbiome samples. Biometrics. 2018 Jun;74(2):448-457. doi: 10.1111/biom.12775. Epub 2017 Oct 9. PMID 28991375